CLINICAL TRIAL: NCT05152004
Title: Efficacies of Hybrid and High-dose Dual Therapies for the First-line Anti-H Pylori Treatment - a Randomized Trial
Brief Title: Efficacies of Hybrid and High-dose Dual Therapies for the First-line Anti-H Pylori Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Chen Tai M.D., Associate professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201800871A3
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori eradication; Hybrid therapy; High dose dual proton pump inhibitor and Amoxicillin therapy
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Interventional Study Model
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose dual therapy (Experimental): Rabeprazole (Pariet) 20 mg and amoxicillin (Amolin) 750 mg q.i.d for 14 days
  Interventions: Drug: Pariet; Drug: Amolin
- Hybrid therapy (Active Comparator): Rabeprazole (Pariet) 20 mg and amoxicillin (Amolin) 1 g b.i.d. for 7 days, followed by rabeprazole (Pariet) 20 mg, amoxicillin(Amolin)1 g, clarithromycin (Klaricid) 500 mg, and metronidazole (Flagyl) 500 mg b.i.d. for 7 days
  Interventions: Drug: Pariet; Drug: Amolin; Drug: Klaricid; Drug: Flagyl

INTERVENTIONS:
Drug: Pariet — Rabeprazole 20 mg and amoxicillin 750 mg qid for 14 days
  Other Names: Rabeprazole
Drug: Amolin — Rabeprazole 20 mg and amoxicillin 750 mg qid for 14 days
  Other Names: Amoxicillin
Drug: Klaricid — Rabeprazole 20 mg and amoxicillin 1 g bid. for 7 days, followed by rabeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg, and metronidazole 500 mg bid. for 7 days
  Other Names: Clarithromycin
  Arms: Hybrid therapy
Drug: Flagyl — Rabeprazole 20 mg and amoxicillin 1 g bid. for 7 days, followed by rabeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg, and metronidazole 500 mg bid. for 7 days
  Other Names: Metronidazole
  Arms: Hybrid therapy

SUMMARY:
Both hybrid and high-dose dual therapies developed by the scholars from Taiwan can achieve a high eradication rate for clarithromycin-resistant strains, and have a great potential to replace bismuth quadruple therapy in the treatment of H. pylori infection. This study aims to better understand the potential of both hybrid and igh-dose dual therapies in the treatment of H. pylori infection.

.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infect more than 50% of humans globally. It is the principal cause of chronic gastritis, gastric ulcer, duodenal ulcer, gastric adenocarcinoma and gastric mucosa-associated lymphoid tissue lymphoma (MALToma). The Real-world Practice & Expectation of Asia-Pacific Physicians and Patients in H. pylori Eradication (REAP-HP) Survey demonstrated that standard triple therapy was still the most commonly used anti-H. pylori regimen in the Asia Pacific region. However, the eradication rates of standard triple therapy have declined to less than 80% in most countries worldwide. The main reasons for eradication failure of standard triple therapy include antibiotic resistance, poor compliance and CYP2C19 genotype of host. Clarithromycin resistance of H. pylori has been identified as the main reason for the failure of standard triple therapy. Pooled data from 20 studies involving 1,975 patients treated with standard triple therapy showed an eradication rate of 88% in clarithromycin-sensitive strains versus 18% in clarithromycin-resistant strains. Therefore, the background rate of clarithromycin resistance is critically important for the efficacy of standard triple therapy. Recently, several strategies including bismuth-containing quadruple therapy, non-bismuth quadruple therapy (i.e., sequential therapy, concomitant therapy and hybrid therapy) and high-dose dual therapy have been proposed to increase the eradication rate.

Hybrid therapy developed by our study group in 2011 consists of a dual therapy with a proton pump inhibitor (PPI) and amoxicillin for 7 days followed by a quadruple regimen with a PPI, amoxicillin, clarithromycin and metronidazole for 7 days [10]. It achieved an eradication rate of 97.4% by intention-to-treat (ITT) analysis and 99.1% by per-protocol (PP) analysis in a Taiwan population with clarithromycin resistance rate of 7%. Subsequent randomized controlled trials demonstrated that 14-day hybrid therapies were comparable or more effective than 10-day sequential therapies. A recent large multicentre randomized controlled trial documented that 14-day hybrid and 14-day concomitant therapies had comparable efficacy in the treatment of H. pylori infection, and both could cure more than 90% of patients with H. pylori infections in areas of high clarithromycin and metronidazole resistance [24]. Therefore, hybrid therapy has a great potential to replace bismuth quadruple therapy in the first-line treatment of H. pylori infection. Currently, hybrid therapy is a recommended first-line treatment for H. pylori infection in the ACG guideline

, Bangkok Consensus Report and Taiwan Consensus Report. High-dose dual therapy developed by Yang et al. is another emerging treatment for H pylori infection. The new therapy consists of high-dose PPI and amoxicillin, which keep the intragastric pH at a value higher than 6.5 regardless of CYP2C19 genotype and maintain steady plasma concentration of amoxicillin above the minimal inhibitory concentration (MIC) for H pylori [28]. The efficacy of the new therapy was significantly higher than that of standard triple therapy in Taiwan. However, it was less effective as the first-line therapy for eradicating H pylori in Korea and in the United States.

This study aims to better understand the potential of both hybrid and igh-dose dual therapies in the treatment of H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. H. pylori-infected outpatients with endoscopically proven peptic ulcer diseases or gastritis.

Exclusion Criteria:

1. Previous H. pylori-eradication therapy
2. ingestion of antibiotics, bismuth, or PPIs within the prior 4 weeks
3. patients with allergic history to the medications used
4. patients with previous gastric surgery
5. the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
6. pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The rates of H.pylori eradication | 4-8 weeks
  The primary outcome variables were the rates of eradication. Chi-square test with or without Yates correction for continuity and Fisher's exact test were used when appropriate to compare the major outcomes between groups. A P value less than 0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Tai, MD, Principal Investigator — Kaohsiung Chang Gung Memorial Hospital,Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Tai WC, Yang SC, Yao CC, Wu CK, Liu AC, Lee CH, Kuo YH, Chuah SK, Liang CM. The Efficacy and Safety of 14-day Rabeprazole Plus Amoxicillin High Dose Dual Therapy by Comparing to 14-day Rabeprazole-Containing Hybrid Therapy for the Naive Helicobacter pylori Infection in Taiwan: A Randomized Controlled Trial. Infect Dis Ther. 2023 May;12(5):1415-1427. doi: 10.1007/s40121-023-00811-3. Epub 2023 May 3. PMID 37133673